CLINICAL TRIAL: NCT00005108
Title: Effects of Hormone Therapy on Vascular Inflammation and Compliance
Brief Title: Effects of Hormone Replacement Therapy on Inflammation and Stiffening of Artery Walls
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 000111; 00-H-0111
Record Dates: First submitted 2000-04-11; First posted 2000-04-12 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-01

CONDITIONS: Atherosclerosis; Healthy; Vascular Disease
Keywords: Menopause; Atherosclerosis; Estrogen; MRI; Ultrasound
MeSH Terms: conditions — Atherosclerosis; Vascular Diseases | interventions — Estradiol; Progesterone

INTERVENTIONS:
Drug: Estradiol
Drug: Progesterone

SUMMARY:
This study will determine the effects of hormone replacement therapy (estrogen alone or estrogen and progesterone) on the walls of arteries in postmenopausal women. Inflammation and stiffness of artery walls are two risk factors for atherosclerosis-deposits of fatty substances (plaques) that can block the vessel, causing a heart attack or stroke. Estrogen raises the levels of certain substances in the blood that cause vessel inflammation and lowers the levels of others. This study will measure the net effects of estrogen on artery wall inflammation and stiffness.

Postmenopausal women in good health may participate in this study. Volunteers will be screened for eligibility with a complete medical history, heart examination, and blood tests. Participants will be randomly assigned to receive either: 1) hormone therapy (estradiol 2 mg daily alone for women who have had a hysterectomy or estradiol plus micronized progesterone 200 mg daily for women with an intact uterus); or 2) placebo (look-alike pills that contain no active drug). Women in both groups will take pills for 3 months, then no pills for 1 month, and then will crossover to the alternate therapy for 3 months (i.e., those in the original placebo group will take hormones, and those in the hormone group will take placebo). At the end of each 3-month treatment period, participants will undergo the following procedures to assess blood vessel inflammation and stiffness:

1. Blood tests - 60 cc (about 2 ounces) of blood will be drawn to measure levels of hormones, cholesterol, and substances in the blood that indicate inflammation of the vessels.
2. Ultrasonography - an ultrasound probe will be applied gently on the neck to image the right and left carotid arteries (arteries in the neck that lead to the brain). During the procedure, the heart's electrical activity will also be monitored with an electrocardiogram and a blood pressure cuff will be wrapped around the arm to obtain blood pressure measurements every 5 minutes.
3. Magnetic resonance imaging (MRI) - Images of the carotid arteries are taken while the volunteer lies on a table in a narrow cylinder containing a magnetic field. A padded sensor called an MRI coil is placed over the neck and earplugs are placed in the ears to muffle the loud noise of the machine during scanning. During the second half of the exam, gadolinium is injected through a catheter (thin, flexible tube) inserted into a vein. Gadolinium is a contrast agent that is used to brighten the scan images.

Information from this study will increase knowledge about the effects of estrogen on vessel wall inflammation. As such, it may be used in the future to help guide decisions about chronic hormone replacement therapy in postmenopausal women.

DETAILED DESCRIPTION:
Vascular inflammation plays an important role in the pathogenesis of atherosclerosis and may contribute to stiffening of arteries that increases the risk of myocardial infarction and stroke. Accordingly, therapies that reduce vascular inflammation may reduce cardiovascular risk. The effect of estrogen therapy on serum markers of inflammation in postmenopausal women is divergent: Estrogen increases the levels of C-reactive protein, interleukin-6, and matrix metalloproteinase-9 ( MMP-9), but decreases levels of the soluble cell adhesion molecules ICAM-1, VCAM-1 and E-selectin. MMP-9 is secreted by macrophages and cytokine-activated smooth muscle cells, with increased expression in the vicinity of atherosclerotic plaques. Although activation of MMP-9 by estrogen could be deleterious in women with coronary artery disease by digesting the fibrous caps of vulnerable plaques and provoking thrombosis (consistent with the Heart and Estrogen/progestin Replacement Study), activation of MMP-9 in healthy postmenopausal women may remove excess matrix proteins that contribute to arterial stiffness (reduced compliance), thus reducing cardiovascular risk (consistent with the Nurses' Health Study). Reduction of levels of cell adhesion molecules might protect against new plaque development in both groups of women. The purposes of this protocol are to determine the net effects of estrogen therapy on 1) vascular inflammation in postmenopausal women, using MRI/MRA imaging of the carotid arteries, and 2) arterial compliance, derived from carotid ultrasonography and blood pressure measurements.

ELIGIBILITY:
Ability to comprehend or unwillingness to sign the consent form.

No use of estrogen therapy within 2 months of this study.

No history of breast cancer, uterine cancer, or estrogen-dependent tumor.

No history of deep vein thrombosis or pulmonary embolus.

No cigarette smokers (within 2 years).

No diabetes mellitus (FBS greater than 120 mg/dL).

Triglycerides less than 400 mg/dL.

Blood pressure less than 160/90 without antihypertensive therapy.

No history of coronary artery disease.

No history of carotid artery disease or stroke.

No history of pancreatitis.

No history of claustrophobia.

No history of involuntary motion disorder.

Specific MRI exclusion criteria (i.e., no pacemaker, no cochlear implants, no AICD, no internal infusion pump, no metal implants or clips in field of view).

No systemic inflammatory disorder (e.g., rheumatoid arthritis, periarteritis nodosa, systemic lupus erythromatosus, temporal arteritis).

Must not have a need for chronic aspirin or NSAID therapy.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 2000-04; Study Completion 2002-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Koh KK, Bui MN, Mincemoyer R, Cannon RO 3rd. Effects of hormone therapy on inflammatory cell adhesion molecules in postmenopausal healthy women. Am J Cardiol. 1997 Dec 1;80(11):1505-7. doi: 10.1016/s0002-9149(97)00732-7. PMID 9399737
- [Background] Cushman M, Legault C, Barrett-Connor E, Stefanick ML, Kessler C, Judd HL, Sakkinen PA, Tracy RP. Effect of postmenopausal hormones on inflammation-sensitive proteins: the Postmenopausal Estrogen/Progestin Interventions (PEPI) Study. Circulation. 1999 Aug 17;100(7):717-22. doi: 10.1161/01.cir.100.7.717. PMID 10449693
- [Background] Hulley S, Grady D, Bush T, Furberg C, Herrington D, Riggs B, Vittinghoff E. Randomized trial of estrogen plus progestin for secondary prevention of coronary heart disease in postmenopausal women. Heart and Estrogen/progestin Replacement Study (HERS) Research Group. JAMA. 1998 Aug 19;280(7):605-13. doi: 10.1001/jama.280.7.605. PMID 9718051